CLINICAL TRIAL: NCT00911391
Title: Prospective, Double-Blinded, Randomised Controlled Trial of Doppler-Optimised Fluid Balance in Elective Colectomy Within an ERAS Protocol
Brief Title: Randomised Trial of Doppler-Optimised Fluid Balance in Elective Colectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Counties Manukau Health (Other); Waitemata District Health Board (Other Government)
Responsible Party: Principal Investigator, SACS, Associate Professor Andrew G Hill, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDFT RCT
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Colorectal Cancer; Colectomy; Surgery; Perioperative Care
Keywords: Doppler; Colectomy; ERAS; Fluid; Perioperative Care
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluid restriction (Active Comparator): Current best practice of intraoperative fluid restriction
  Interventions: Procedure: Intraoperative fluid restriction
- Oesophageal Doppler (Experimental): Oesophageal Doppler-guided fluid administration
  Interventions: Device: Oesophageal Doppler

INTERVENTIONS:
Device: Oesophageal Doppler — Non-invasive measurement of doppler-derived cardiovascular variables (CO, aortic flow rate). Used safely over 800, 000 times
  Other Names: CardioQ Deltex Oesophageal Doppler
  Arms: Oesophageal Doppler
Procedure: Intraoperative fluid restriction — Current best practice of avoiding fluid overload by intraoperative fluid restriction
  Arms: Fluid restriction

SUMMARY:
Perioperative fluid management has been historically dictated by outdated, contradictory concepts. Excessive or inadequate fluid administration around surgery is deleterious and hence goal-directed fluid therapy using Oesophageal Doppler-derived cardiac indices is preferable to optimize tissue perfusion. Previous studies in this area have been hampered by lack of standardization in other aspects of perioperative care and none have explored the impact of individualized fluid therapy on post-operative fatigue.The investigators proposed a study involving 80 patients having open/ laparoscopic colonic surgery to investigate the effect of Oesophageal Doppler guided fluid administration intraoperatively compared to current best practice of fluid restriction. The investigators have an optimized peri-operative care pathway established at the Manukau Surgical Centre (MSC), Middlemore Hospital. All patients will be cared for under the Enhanced Recovery After Surgery (ERAS) multimodal care plan therefore ensuring that all other aspects of care besides intraoperative fluid administration remain homogenous. Outcomes will include post-operative recovery, clinical outcomes as well as physiological data with follow-up to 30 days.

DETAILED DESCRIPTION:
Until very recently, modern perioperative fluid management has involved routine administration of large quantities of fluids during major surgical procedures, typically causing a weight increase of 3-6 kg in the early post-operative period.Several factors, including concern about preoperative dehydration, attempts to support the circulation and cardiac function after general and regional anaesthesia, prevention of blood transfusion and maintenance of adequate kidney perfusion have historically lead to excess perioperative fluid administration.

However administration of excess fluid has been shown to contribute to postoperative morbidity. It increases demand on the heart and may adversely affect postoperative cardiac function. It may also lead to increased pulmonary complications. Fluid overload may lead to oedema of the gastrointestinal tract and hence contribute to post-operative gastrointestinal paralysis, bacterial translocation and sepsis. Excess fluid also has been shown to decrease tissue oxygen tension with potential deleterious effects on anastomotic and wound healing.

Therefore, current best practice has centred on fluid restriction peri-operatively with an increased focus on the intraoperative fluid regimen. Since hypovolaemia is also associated with a myriad of adverse outcomes, a balanced perioperative intravenous fluid regimen focussing on tissue perfusion is thought to be optimal. By using the Oesophageal Doppler Monitor (ODM) as a means to non-invasively estimate intra-operative cardiac output, significant improvements in outcome have been observed in patients undergoing major orthopaedic and cardiac procedures. Previous studies in patients undergoing major abdominal surgery have demonstrated that goal-directed intraoperative fluid administration using ODM may result in improved outcomes such as reduced number of critical care admissions, reduced hospital stay and overall decreased morbidity.

In the broader context of perioperative care in colonic surgery, recent developments have included Enhanced Recovery After Surgery (ERAS) programmes- a combination of various evidence-based strategies implemented together as part of a standardised protocol to synergistically decrease post-operative fatigue and improve outcomes. These strategies include preoperative counselling, avoidance of mechanical bowel preparation, pre-operative carbohydrate loading, perioperative high-flow oxygen therapy, mid-thoracic epidural analgesia, avoidance of parenteral opioids and routine wound drainage, use of short or transverse incisions, early mobilisation, early feeding and a balanced analgesia regiment. ERAS protocols are also ideal for well-designed clinical trials as they provide a template to trial new interventions on the background of an otherwise homogenous, optimised perioperative care programme. An ERAS programme has been implemented and prospectively evaluated at Manukau Surgical Centre, Middlemore Hospital in Auckland.

In a recently published systematic review, we identified that a major short-coming of the literature in this field is the non-standardised nature of peri-operative management of the patients in these studies. Although fluid management was optimised, the other aspects of care were not optimised or even standardised, introducing the risk of significant confounding. Furthermore, none have explored the role of fluid management on post-operative functional recovery- an important metric of patient-relevant outcomes evaluating recovery beyond physiological and clinical parameters. Furthermore, none of the published ERAS programmes have used ODM as part of their peri-operative strategies. Consequently, the true impact of optimised fluid therapy within an environment of current best-practice (ERAS) is unknown.

Methods Research Design We will conduct a double-blinded, randomised controlled trial of ODM versus fluid restriction (current best-practice) in patients undergoing colonic surgery within our ERAS programme to determine whether individualising fluid administration enhances post-operative recovery, thereby improving patient outcomes.

Sample Size:

To detect a 20% improvement in recovery as measured by the Surgical recovery Score at Day 7 (based on data from our previous work), we will require 37 patients in each arm (α= 0.05, β= 0.8) Therefore, we shall aim to recruit 80 patients anticipating for possible drop-outs.

Patients will be consented and then randomised by computer generated random numbers and the opaque envelope method. All Patients will have an oesophageal probe inserted with readings not available to the anaesthetist for patients in the control group (the screen will be covered). At the commencement of anaesthesia, the patient will be randomised to receive fluid management optimised by ODM data or by standard parameters. The patients, surgeons and investigators will be blinded to the intervention. The anaesthetists will use a validated protocol for the treatment group. Measurements of cardiac indices (Cardiac Output, Aortic Flow Rate) from the ODM will be noted intraoperatively. The Oesophageal probe shall be removed at the end of surgery prior to the patient waking up. All other aspects of perioperative care will be according to our previously developed ERAS programme.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients undergoing open/ laparoscopic colonic resection at Manukau surgical Centre (MSC)or North Shore Hospital, Auckland.

Exclusion Criteria:

* severe oesophageal disease
* recent oesophageal or upper airway surgery
* moderate or severe aortic valve disease as proven by echocardiogram
* documented bleeding diathesis
* preoperative steroid use
* cognitive impairment
* ASA>3
* patient choice.
* rectal tumour (defined as less an 15cm from anal verge on preop investigations)
* creation of stoma
* difficulty in obtaining reliable measurements from ODM

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2009-11; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Post-operative functional recovery | 7 day

SECONDARY OUTCOMES:
Perioperative Complications | 30 day
  As defined using trial by Buzby et al Am J Nutr 1989 and graded according to Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Hill, MBChB MD FRACS, Principal Investigator — South Auckland Clinical School, University of Auckland
Locations (2):
- New Zealand (2):
  - Manukau Surgery Centre-Middlemore Hospital, Auckland, Auckland
  - North Shore Hospital, Auckland

REFERENCES:
- [Derived] Srinivasa S, Taylor MH, Singh PP, Yu TC, Soop M, Hill AG. Randomized clinical trial of goal-directed fluid therapy within an enhanced recovery protocol for elective colectomy. Br J Surg. 2013 Jan;100(1):66-74. doi: 10.1002/bjs.8940. Epub 2012 Nov 6. PMID 23132508